CLINICAL TRIAL: NCT00881699
Title: Randomized Clinical Trial of a Brazilian HIV Prevention Intervention for the Severely Mentally Ill
Brief Title: Testing an HIV Prevention Intervention for Psychiatric Patients in Brazil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #5264; R01MH065163 (NIH); DAHBR 9A-ASPI
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infection; HIV Infections
Keywords: HIV Information; HIV Prevention; Severe Mental Illness; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will complete HIV risk reduction group meetings.
  Interventions: Behavioral: HIV Prevention Intervention - Project PRISSMA - HIV I have my eye on you
- 2 (Active Comparator): Participants will complete health promotion group meetings.
  Interventions: Behavioral: Health Promotion Intervention

INTERVENTIONS:
Behavioral: HIV Prevention Intervention - Project PRISSMA - HIV I have my eye on you — Eight weekly 2-hour HIV risk reduction intervention sessions, with three weekly 2-hour booster sessions completed 6 months after the initial intervention. Specific goals of the intervention are to (1) increase information about HIV risk behaviors and safer sex options; (2) increase identification of personal risk of HIV and enhance the motivation to engage in safer sex behaviors; and (3) enhance skills to achieve safer sex, particularly negotiating safer sex, using condoms, and communicating within a relationship.
  Arms: 1
Behavioral: Health Promotion Intervention — Eight weekly 2-hour health promotion intervention sessions with three weekly 2-hour booster sessions completed 6 months after the initial intervention. Specific goals of the intervention are to (1) increase information about health issues specific to psychiatric patients, (2) increase identification of personal health risks and enhance motivation to engage in healthier behaviors, and (3) enhance skills to achieve healthier behaviors.
  Arms: 2

SUMMARY:
This study will test the effectiveness of a program aimed at reducing behaviors that increase HIV risk among people with severe mental illnesses.

DETAILED DESCRIPTION:
HIV is a virus that weakens a person's immune system and can cause AIDS. It is most commonly transmitted through unprotected sexual contact. People with a mental illness who are sexually active may be at risk of HIV infection, but most interventions for reducing risk of HIV infection do not target this particular population. This study will test an intervention aimed at reducing behaviors with a high risk of causing HIV infection in sexually active people with a mental illness.

Participation in this study will last 15 months. At study entry, participants will complete a baseline interview with a research assistant. This interview will evaluate sexual activity, knowledge of HIV, the participant's psychiatric diagnosis and symptoms, attitude toward condoms, and stigma related to mental illness experienced by the participant.

Participants will then be randomly assigned to either an HIV risk reduction group or a general health group. Both of these groups will meet once a week for 8 weeks. Those in the HIV risk reduction group will learn information and take part in activities aimed at reducing behaviors that place people at a high risk of being infected with HIV. Those in the general health group will learn about long-term serious medical conditions, such as diabetes and high blood pressure, that may be common in people with a mental illness.

Participants will complete two follow-up visits after their 8-week intervention, one the week after and one 3 months after. Participants will then complete a "booster" of three weekly group sessions covering the same information from their 8-week intervention. More follow-up visits will occur 1 week and 6 months after participants complete the booster sessions. All follow-up visits will involve an interview similar to the one held at study entry. Additionally, feedback forms will be completed at the first interview at study entry, after the eight group sessions, after the three booster sessions, and at the last interview.

ELIGIBILITY:
Inclusion Criteria:

* Being treated as a patient in one of the study psychiatric clinics
* Sexually active in the past 3 months

Exclusion Criteria:

* Primary alcohol or other drug use disorder
* Acutely psychotic or actively suicidal at the time of the screening interview
* Developmental disability as a primary diagnosis
* Unable to speak Portuguese

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2006-09; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sexual Risk Behavior Assessment Schedule (SERBAS) | Measured at baseline and 3, 6, and 12 months post-intervention

SECONDARY OUTCOMES:
Brief HIV Knowledge Questionnaire (Brief HIV-KQ) | Measured at baseline and 3, 6, and 12 months post-intervention
Brief Psychiatric Rating Scale (BPRS) | Measured at baseline and 3, 6, and 12 months post-intervention
Stigma and Discrimination Questionnaire | Measured at baseline and 3, 6, and 12 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Milton L. Wainberg, MD, Principal Investigator — Columbia University and New York State Psychiatric Institute
Locations (1):
- Instituto de Psiquiatria da Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Wainberg ML, Mann CG, Norcini-Pala A, McKinnon K, Pinto D, Pinho V, Cavalcanti MT, Cheng-Shiun L, Guimaraes MD, Mattos P, Hughes E, Palinkas LA, Otto-Salaj L, Remien RH, Cournos F. Challenges and opportunities in the science of research to practice: lessons learned from a randomized controlled trial of a sexual risk-reduction intervention for psychiatric patients in a public mental health system. Braz J Psychiatry. 2020 Aug;42(4):349-359. doi: 10.1590/1516-4446-2019-0737. Epub 2020 Jan 24. PMID 31994641